CLINICAL TRIAL: NCT00488371
Title: Evaluation of Streptococcus Pneumoniae Nasopharyngeal Carriage Rate in Children Receiving Pneumococcal Conjugated Vaccine (Prevnar®) Under the Auspices of the Taipei City Government Vaccination Program
Brief Title: Study Evaluating Streptococcus Pneumoniae Nasopharyngeal Carriage Rate in Children Receiving Prevnar®
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0887X1-4410
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2007-12-20 (Estimated); Status verified 2007-12

CONDITIONS: Pneumococcal Infections
Keywords: Streptococcus pneumoniae nasopharyngeal carriage
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Pneumococcal Conjugated Vaccine (Prevnar®)

SUMMARY:
Primary Objective:

To evaluate the impact of PCV7 vaccination on NP carriage rate of vaccine serotypes and serotype distribution

Secondary Objective:

To evaluate the impact of PCV7 vaccination on NP carriage of antibiotic resistant pneumococci and serotype distribution.

DETAILED DESCRIPTION:
Under the Social Welfare Vaccination Program, the Taipei City Government will vaccinate approximately 5,000 children residing in the city of Taipei between 2 and 5 years of age during the months of November 2006 to April 2007 with one dose of PCV7.

To gather baseline data on serotype distribution and antibiotic resistance of nasopharyngeal (NP) carriage isolates in this population and measure vaccine impact on NP carriage, the Taipei city government requires the evaluation of the vaccination program through the detection of Streptococcus pneumoniae NP carriage rate pre and post vaccination in a convenience sample of approximately 1000 children. This number complies with the Taipei city government request for the inclusion of 250 children.

Streptococcus pneumoniae is a major cause of bacterial otitis media, pneumonia, sepsis, bacteraemia, and meningitis among infants worldwide.

The main reservoir of pneumococci is the human nasopharynx. The mean age of first acquisition is 6 months and carriage rates peak in the preschool age group. The organisms have pilli on their surface to assist in adhering to nasopharyngeal mucosal receptors. Streptococcus pneumoniae is part of the normal flora in colonized individuals, but the organism has the ability to cause disease by invading neighboring tissues, and potentially spreading into the bloodstream and other sites, causing invasive pneumococcal disease, such as bacteremia, sepsis and meningitis. The rate of NP carriage for Streptococcus pneumoniae in Taiwan (1998-99) was estimated to be 19.9 % overall for children 1-14 years and 27.1 % for those 2-5 years. A more recent study by Lauderdale et al. found a carriage rate of 41 % in children attending a kindergarten program in Taiwan where a 5 year old was diagnosed with streptococcus meningitis.

Prevnar® has shown a high degree of efficacy in the prevention of invasive pneumococcal disease in children. In addition, PCV7 has been shown to decrease NP carriage of serotypes included in the vaccine (VST). Since NP carriage is a prerequisite for transmission of Streptococcus pneumoniae, decrease in NP carriage of VSTs in children has resulted in decreased transmission to their contacts and an indirect effect (herd effect) on invasive pneumococcal disease. Since the majority of antibiotic resistant strains are VST, PCV7 immunization has decreased antibiotic resistance in invasive pneumococcal disease for both those immunized and their contacts. However, after PCV7 vaccination overall pneumococcal NP carriage rates do not change, since Streptococcus pneumoniae serotypes not included in the vaccine (NVST) replace the VSTs. Although in the nasopharynx there is an almost complete replacement by NVST, these serotypes may have less ability to cause invasive disease, since disease with NVST has been observed but to a much lower magnitude than disease prior to PCV7 vaccination.

Thus, the expected outcome of a successful PCV7 vaccination program on NP carriage is a decrease in carriage of VST with an increase in NVST and thus, a stable overall Streptococcus pneumoniae carriage rate.

ELIGIBILITY:
Inclusion criteria

* Healthy children aged 2 to 5 years old identified by the Taipei City government and are participating in Taipei City's PCV7 vaccination program.
* Informed consent obtained from parents or legal guardian.
* Eligible to receive 1 dose of PCV7

Exclusion criteria

* Children with any of the following conditions: immunologic diseases; neoplastic disorders; renal, cardiac, hepatic, or hematologic diseases; bronchodysplasia; Down syndrome; chronic otitis media with effusion.
* Children with any acute illness including mild acute respiratory infection or fever > 38 centigrade.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250
Dates: Start 2006-11; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Taiwan, medinfo@wyeth.com